CLINICAL TRIAL: NCT05368038
Title: ScreenPlus: A Comprehensive, Flexible, Multi-disorder Newborn Screening Program
Acronym: ScreenPlus
Status: Enrolling by invitation | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Alexion Pharmaceuticals, Inc. (Industry); BioMarin Pharmaceutical (Industry); Cure Sanfilippo Foundation (Unknown); Dana's Angels Research Trust (DART) (Unknown); Mirum Pharmaceuticals, Inc. (Industry); Orchard Therapeutics (Industry); Passage Bio, Inc. (Industry); Genzyme, a Sanofi Company (Industry); Sio Gene Therapies (Industry); Takeda Pharmaceuticals North America, Inc. (Industry); The FireFly Fund (Unknown); The Noah's Hope - Hope 4 Bridget Family Foundations (Unknown); Travere Therapeutics, Inc. (Industry); Ultragenyx Pharmaceutical Inc (Industry); Ara Parseghian Medical Research Fund (Unknown); New York State Department of Health (Other Government); Case Western Reserve University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-10774; R01HD073292 (NIH)
Record Dates: First submitted 2022-04-06; First posted 2022-05-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Acid Sphingomyelinase Deficiency; Ceroid Lipofuscinosis, Neuronal, 2; Cerebrotendinous Xanthomatosis; Fabry Disease; GM1 Gangliosidosis; Gaucher Disease; Lysosomal Acid Lipase Deficiency; Metachromatic Leukodystrophy; Mucopolysaccharidosis II; Mucopolysaccharidosis III-B; Mucopolysaccharidosis IV A; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Niemann-Pick Disease, Type C
Keywords: Newborn Screening; Rare Diseases; Families; Genetics; ELSI
MeSH Terms: conditions — Niemann-Pick Diseases; Ceroid Lipofuscinosis, Neuronal, 2; Xanthomatosis, Cerebrotendinous; Fabry Disease; Gangliosidosis, GM1; Gaucher Disease; Wolman Disease; Leukodystrophy, Metachromatic; Mucopolysaccharidosis II; Mucopolysaccharidosis III; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Niemann-Pick Disease, Type C; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn infants born at a ScreenPlus pilot hospital: Parents who give permission will have their infant's sample screened for the ScreenPlus panel. Infants who screen positive after multi-tiered testing will be referred to a ScreenPlus doctor for confirmatory testing and care coordination.
  Interventions: Diagnostic Test: Confirmatory Testing

INTERVENTIONS:
Diagnostic Test: Confirmatory Testing — All positive screens will be referred using standard notification procedures, where the New York State NBS reporting team contacts the ScreenPlus site medical geneticist, who will contact the newborn's pediatrician and family. The initial evaluation will include a clinical examination and confirmatory molecular studies, enzymatic and biomarker studies, when available. All aspects of the confirmatory testing will be at no cost to the participants. If confirmed to have a ScreenPlus disorder, the investigators will counsel the family and help connect them with treatment, clinical trials and disease specialists. The investigators will also provide emotional and social support resources to help in this journey.

SUMMARY:
ScreenPlus is a consented, multi-disorder pilot newborn screening program implemented in conjunction with the New York State Newborn Screening Program that provides families the option to have their newborn(s) screened for a panel of additional conditions. The study has three primary objectives: 1) define the analytic and clinical validity of multi-tiered screening assays for a flexible panel of disorders, 2) determine disease incidence in a large newborn population, and 3) assess the impact of early diagnosis on health outcomes. Over a nine-year period, ScreenPlus aims to screen 100,000 infants born in eight high birthrate hospitals in New York for a flexible panel of rare genetic disorders. This study will also evaluate the Ethical, Legal and Social issues pertaining to NBS for complex disorders, which will be done via online surveys that will be directed towards ScreenPlus parents who opt to participate and qualitative interviews with families of infants who are identified through ScreenPlus.

DETAILED DESCRIPTION:
Soon after birth, all babies born in the United States have a newborn screening (NBS) test to check for certain medical conditions. All babies are screened, even if they appear healthy, because most of these conditions have no obvious physical findings in a newborn and might otherwise be diagnosed only after the development of serious problems, such as brain damage, organ damage, or death. In fact, NBS has been an integral part of preventable health care for over five decades, ever since the discovery that phenylketonuria is an easily diagnosed, preventable cause of intellectual disability.

Over the past two decades, there have been dramatic advances in screening technology, with a resulting increase in the number and complexity of disorders on NBS panels. This enhanced ability to screen brings questions about what types of disorders are appropriate for NBS. To that end, the Advisory Committee on Heritable Disorders in Newborns and Children (ACHDNC) was established in 2003 to make evidence-based recommendations at the national level regarding the suitability of various disorders for NBS. At present, the Recommended Uniform Screening Panel (RUSP) includes 35 core disorders. The RUSP nomination process uses information about disease incidence and severity, natural history, benefits of early detection, safety and efficacy of treatment, analytic and clinical validity of the screening tests, as well as consideration of potential harms associated with screening and public health impact to determine whether a particular disorder is appropriate for NBS. However, there are many disorders for which this data is insufficient or missing. There are other disorders that challenge traditional NBS criteria by having predominantly later-onset phenotypes, poorly defined natural history, or unclear treatment outcomes. As these potentially life-threatening disorders might benefit from early detection, gathering and analyzing this data is both critical and timely. Accordingly, there is a great deal of interest in pilot NBS studies as a means to gather objective evidence about whether a disorder is appropriate for widespread screening.

ScreenPlus is a comprehensive, fluid, pilot NBS program that will screen 100,000 consented infants for specific disorders that are under consideration for universal NBS. This study will generate critical data about the validity of testing for these candidate disorders and provide estimates of disease incidence in a large newborn population. The investigators will evaluate different consent and engagement models, including direct, in-person interaction and the use of an electronic consent framework to educate parents about pilot NBS. The investigators will also collect nuanced information about the ethical implications of NBS, by conducting qualitative interviews with parents of children who have received a positive or uncertain NBS result. Parents who are eligible to participate in ScreenPlus will also have the opportunity to complete a flexible set of surveys of parent opinions about expanded NBS, research using dried blood spots, and other relevant topics. Furthermore, newborns who screen positive will be followed by a ScreenPlus physician. Through thoughtful collaboration with disease experts, the investigators will help systematically collect disease specific measures through detailed long-term follow-up which will enable us to critically evaluate how affected children identified through ScreenPlus are faring, allowing objective assessment of the impact early diagnosis has on outcome.

The investigators will share this important data with the NBS community to help inform objective decision-making about widespread screening recommendations. The ScreenPlus panel is fluid and disorders may be added/removed as disorders satisfy the study inclusion criteria. Additionally, recognizing that the NIH, advocacy groups, academics, and private industry all share a desire for clean, consented pilot NBS data, the investigators created a unique financial infrastructure. This investigator-driven arrangement permits all stakeholders to obtain aggregate data of interest in a mutually beneficial and cost-effective manner. ScreenPlus is guided by Scientific and Community Advisory Boards, who are comprised of rare disease experts, biochemistry specialists, physicians, bioethicists, and patient advocates. Overall, the investigators anticipate that ScreenPlus will become the premier consented pilot NBS program in the United States.

In sum, ScreenPlus will provide critical data about the appropriateness of NBS for candidate disorders, the feasibility and effectiveness of consented screening models, and parent informational needs and preferences as they relate to NBS for complex disorders.

ELIGIBILITY:
Inclusion Criteria:

* All newborn infants born at a ScreenPlus pilot hospital
* Infants who are less than four weeks old, regardless of sex, gestational age, or health status.

Exclusion Criteria:

* A newborn screening sample is unavailable
* Infants who are more than four weeks old

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns born at a ScreenPlus pilot hospital who are less than four weeks old.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the accuracy of the screening assays. | Through study completion up to 9 years.
  Accuracy of the screening assay will be defined in terms of positive predictive value (proportion of confirmed cases comparative to the total number of infants who screened positive).
Define disease incidence in a large newborn population. | Through study completion up to 9 years.
  Disease incidence will be calculated as the proportion of infants with a disorder comparative to the total population of infants screened.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Wasserstein, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (9):
- United States (9):
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Health - Tisch Hospital, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Long Island Jewish Medical Center, Queens, New York
  - Jack D. Weiler Hospital, The Bronx, New York
  - ScreenPlus Coordinating Core, Children's Hospital at Montefiore, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly NR, Orsini JJ, Goldenberg AJ, Mulrooney NS, Boychuk NA, Clarke MJ, Paleologos K, Martin MM, McNeight H, Caggana M, Bailey SM, Eiland LR, Ganesh J, Kupchik G, Lumba R, Nafday S, Stroustrup A, Gelb MH, Wasserstein MP. ScreenPlus: A comprehensive, multi-disorder newborn screening program. Mol Genet Metab Rep. 2023 Dec 14;38:101037. doi: 10.1016/j.ymgmr.2023.101037. eCollection 2024 Mar. PMID 38173711
- [Background] Calonge N, Green NS, Rinaldo P, Lloyd-Puryear M, Dougherty D, Boyle C, Watson M, Trotter T, Terry SF, Howell RR; Advisory Committee on Heritable Disorders in Newborns and Children. Committee report: Method for evaluating conditions nominated for population-based screening of newborns and children. Genet Med. 2010 Mar;12(3):153-9. doi: 10.1097/GIM.0b013e3181d2af04. PMID 20154628
- [Background] Wasserstein MP, Caggana M, Bailey SM, Desnick RJ, Edelmann L, Estrella L, Holzman I, Kelly NR, Kornreich R, Kupchik SG, Martin M, Nafday SM, Wasserman R, Yang A, Yu C, Orsini JJ. The New York pilot newborn screening program for lysosomal storage diseases: Report of the First 65,000 Infants. Genet Med. 2019 Mar;21(3):631-640. doi: 10.1038/s41436-018-0129-y. Epub 2018 Aug 10. PMID 30093709
- See also: Official ScreenPlus information page on the Albert Einstein College of Medicine website. — https://einsteinmed.edu/research/screenplus/